CLINICAL TRIAL: NCT01239225
Title: Prevalence of Abdominal Aortic Aneurysm in Patients Undergoing Coronary Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Dr. Kyryl Derkach, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: mmc2010137-09ctil
Record Dates: First submitted 2010-11-07; First posted 2010-11-11 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2010-10

CONDITIONS: Coronary Angiography
Keywords: Patients undergoing coronary angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abdominal ultrasound (Experimental): Abdominal ultrasound
  Interventions: Device: Abdominal ultra-sound; Procedure: Abdominal ultrasound

INTERVENTIONS:
Device: Abdominal ultra-sound
Procedure: Abdominal ultrasound

SUMMARY:
Abdominal aortic aneurysms (AAA) are localized, blood-filled dilations (balloon-like bulges) of the aorta. Approximately 90% of abdominal aortic aneurysms occur infrarenally (1). It is most commonly asymptomatic and can be detected randomly during screening. Its prevalence rate in men aged 65 years and more is 5 - 8% (3).

The risk factors for the occurrence of AAA are male gender, advanced age, history of atherosclerosis, cigarette smoking and 1st degree family history (4).

The prevalence rate is higher in patients with history of atherosclerosis of peripheral blood vessels and coronary arteries (5 - 7). As the size of an aneurysm increases, there is an increased risk of rupture, which can result in severe hemorrhage and death. The death rate due to rupture in the elderly population is 90% (3, 8). Elective surgical repair of the abdominal aortic aneurysm is associated with a death rate of 8% (9). Therefore, the importance of the screening of populations at elevated risk is obvious (5 - 7, 10 -14). Among imaging techniques, ultrasonographic screening for abdominal aortic aneurysm is technically simple, accurate and devoid of ionizing radiation. Ultrasonographic diagnosis of AAA is associated with a major reduction in the incidence of abdominal aortic aneurysm-related mortality (15 - 19). The sensitivity of ultrasonographic screening for abdominal aortic aneurysm is about 100% (19). The most common clinical indications for ultrasonographic screening for abdominal aortic aneurysm are a palpable abdominal mass, hemodynamic impairment of aortic system in lower extremities, pain in the chest, lower back or scrotum, and abdominal bruits.

Ultrasonography is used to screen for aneurysms when the outer aortic diameter is more than 3 cm (normal diameter of the aorta is around 2 cm (20). There is disagreement regarding the follow-up of patients after detection of abdominal aortic aneurysm in diameter of 2.6 cm - 2.9 cm (22). Random detection of abdominal aortic aneurysm where the aortic diameter is 2.6 cm, in men aged 65 years and more, have been associated with no risk for its future significant development (21). Ultrasonographic evaluation of abdominal aorta is a challenge for clinicians because of the need for the accurate detection of aortic diameter (20).

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age.
* Subject understands study requirements and diagnostic procedures and agrees to sign an informed consent form prior to both study procedures:

  * Ultrasonographic screening of abdominal aorta (from diaphragm to aorta bifurcation) in horizontal and vertical position for the detection of aneurysms. Ultrasonographic screening will be perform in frontal technique for sagital view and in right lateral decubitus for coronal view. The outer aortic diameter will be measured in three levels: at the level of the diaphragm, at SMA level and proximal to the aorta bifurcation.
  * Coronary angiography.
* The patients will be divided into two groups according to the results of their angiograms:

  * Normal coronary angiography (n=100).
  * Atherosclerosis of coronary arteries (n=100).
  * Subject will be available for ultrasonographic follow-up after the procedure.

Exclusion Criteria:

* Pregnancy.
* Subject has systemic infection, or is suspected of having systemic infection.
* Subject has an untreatable bleeding.
* Enrollment in another study protocol.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual)